CLINICAL TRIAL: NCT03307473
Title: Total Physical Activity and Sedentary Behaviour Changes Associated With Regular Daily Life Utilitarian E-bike Use : VELONAPS Study
Brief Title: Physical Activity and Sedentary Behaviour Associated With Utilitarian E-bike Use
Acronym: VELONAPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: ONAPS : Observatoire National de l'Activité Physique et de la Sédentarité (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-354
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2019-03

CONDITIONS: All-comers
Keywords: Physical activity; Bicycling; Transportation; Public health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- e-bike: During 3 months in a the geographic area of Clermont-Ferrand (France), new e-bike buyers and renters are invited to take part in VELONAPS study before starting to use their e-bike
  Interventions: Behavioral: E6BIKE

INTERVENTIONS:
Behavioral: E6BIKE — During 3 months in a the geographic area of Clermont-Ferrand (France), new e-bike buyers and renters are invited to take part in VELONAPS study before starting to use their e-bike

SUMMARY:
Physical inactivity and sedentary are recognized as important risks factors for several diseases and total mortality. One of the main perceived barriers to physical activity is the lack of time and motivation. Active commuting during daily routine could overcome these barriers and e-bikes appears to be a promising and practical tool to meet physical activity guidelines.

E-bikes are a physically active transportation mode, with a riding intensity contributing to activities in the moderate-intensity range (3-6 METs) for any of the assistance mode. Electric assistance is provided only when a rider is pedaling. The study VELONAPS mainly aims at investigating if real-life usage of utilitarian e-bike is associated with significant changes on total physical activity and sedentary patterns. During up to 4 months of free use of an e-bike, our purpose is to quantify its usage along with total physical activity and sedentary levels. We hypothesize that using an e-bike for commuting increase the total physical activity of at least 7.5 MET-h/week, increasing as well adherence to physical activity guidelines.

DETAILED DESCRIPTION:
During 3 months in a the geographic area of Clermont-Ferrand (France), new e-bike buyers and renters are invited to take part in VELONAPS study before starting to use their e-bike. The sample is constituted of willing participants who plan to use their e-bike, at least in part, for work-related and commuter trips. Each participant will be followed during 4 months, with 4 study points.

At T0, subjects are invited for the baseline visit including a medical interview and physical examination (with anthropometric measurements), and a physical stress test evaluating aerobic fitness (submaximal step-test). Online questionnaires are provided to measure physical activity and sedentary patterns (RPAQ), motivations and barriers to physical activity (EMAPS and BPAQ), perceived health and quality of life (SF-12), perceived exertion for common physical efforts (Borg scale).

At T1 and T2 (respectively one and two months after having started e-bike use), the questionnaire measuring physical activity and sedentary patterns of the past month is requested again.

At T4 (final study point, after 4 months of e-bike use), subjects are invited for the follow-up visit including anthropometric measurements and a physical stress test evaluating aerobic fitness. Online questionnaires are provided to measure the same dimensions than at the T0 study point.

The primary endpoint of the study is to compare the physical activity level at T0 and the one at T4.

Secondary endpoints are the modifications (comparisons between T0 and T4) in :

* sedentary levels.
* the percent of individuals meeting the physical activity guidelines.
* motivations and barriers to physical activity.
* perceived health and quality of life.
* perceived exertion for common physical efforts.
* anthropometric measurements (BMI and waist size). Subgroup analyses will identify either consistency of, of large differences, in the magnitude of e-bike use effect among different categories of participants: by age, by sex, by initial physical condition, and by initial total physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* being a new e-bikes user
* planning to use the e-bikes, at least in part, for work-related and commuter trips

Exclusion Criteria:

* having used regularly (more than once a week) an e-bike for at least one month during the last three months
* e-bike use already started for more than a week
* e-bike use only for leisure activities (no commuting)
* health condition(s) contraindicating a fitness test
* being pregnant
* not having access to the e-bike for a long period (> 1 month) during the follow-up study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: new e-bikes user
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Total physical activity | at 4 months
  the amount of total physical activity engaged in each week (in MET-h/week).

SECONDARY OUTCOMES:
Sedentary time | at 4 months
  Total of time while sitting, lying down, and expending very little energy (approximately 1.0-1.5 metabolic equivalents [METs]) in each day (in h/day).
Physical condition | at 4 months
  Estimated aerobic fitness (in METs)
Exercise motivations questionnaire | at 4 months
  factor structure examination of the Behavioural Regulation in exercise questionnaire-2 (BREQ-2)
Quality of life questionnaire | at 4 months
  Assessment of health related quality of life using SF-12 questionnaire
Weight | at 4 months
  Body weight
Waist size | at 4 months
  Waist size measurement (between the last/lowest rib, and the hip bone)
Perceived exertion | at 4 months
  Rating of perceived exertion for common physical stresses.

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France